CLINICAL TRIAL: NCT05013346
Title: Understanding the Characteristics of Young-onset Diabetes in Sub-Saharan Africa
Brief Title: Characteristics of Young-onset Diabetes in Sub-Saharan Africa (YODA) Study
Acronym: YODA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: University of Yaounde 1 (Other); University of Exeter (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor, Yaounde Central Hospital
Other Study IDs: CNO012021
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes; Diabetes, Autoimmune
Keywords: Type 1 diabetes, C-peptide, islet auto-antibody, sub-Saharan Africa
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva: 2ml of saliva sample will be provided into a saliva pot (GeneFix Saliva Tube Collector) which will be stored at ambient temperature and shipped to the University of Exeter Medical School where DNA will be extracted and analysed.
  Whole Blood: 5ml of whole blood will be collected to be used directly for full blood count and A1c determination.
  Plasma: 10ml of whole blood will be collected into an EDTA tube which will be centrifuged and aliquoted into four (4) 1.8mL cryotubes and stored immediately at minus 80 degrees Celsius pending batch analysis.
  Serum: 10ml of whole blood will be collected into a plain tube which will be centrifuged and aliquoted into four (4) 1.8mL cryotubes and stored pending batch analysis.
  Urine: 10ml of Urine will be collected into a urine collection pot, dipstick urinalysis will be performed immediately and 1.8mL of urine will be stored pending batch analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention needed — No intervention required. Not a clinical trial

SUMMARY:
Type 1 diabetes has been poorly characterised, with very sparse information available in the literature about the characteristics of the disease in Africa. Atypical young onset diabetes is often reported by clinicians in sub-Saharan Africa, including patients who have the phenotype of type 1 diabetes but do not appear to have an absolute insulin requirement. The onset of type 1 diabetes in many sub-Saharan African populations seem to occur at later ages (20s to 40s) than what is generally seen in Caucasian populations. The investigators seek to characterise young-onset insulin treated diabetes (clinically diagnosed type 1 diabetes) in sub-Saharan Africa;

DETAILED DESCRIPTION:
The specific objectives will be to; (1) characterise a population with clinically diagnosed type 1 diabetes and to determine the proportion of islet autoantibody positivity rates and to compare with a similar cohort of patients in the UK, (2) to determine the proportion of participants with retained endogenous insulin secretion (C-peptide > 600pmol/l) and whether they have evidence of autoimmunity as assessed by islet autoantibody and the type 1 diabetes genetic risk score

Study setting: This study will be a multi-center cross-sectional study of clinically diagnosed type 1 diabetes patients who are currently on insulin treatment who are being followed-up in existing diabetes care centers in 4 sub-Saharan African countries; Cameroon, Uganda, Tanzania and South Africa. Recruitment will take place at regional diabetes care centers which usually serve as the main diabetes treatment hub for many smaller spoke clinics in the sub-region. In Cameroon, the Yaounde Central Hospital and the Bafoussam Regional Hospital will serve as main clinical sites. In Uganda the clinical sites involved are the Mulago National Referral and Teaching Hospital, St. Francis Hospital Nsambya, all in Kampala and the Masaka Regional Referral Hospital. The Muhimbili National Hospital in Dar Es Salaam will serve as the main clinical site in Tanzania. Cameroon, Uganda and Tanzania will carry out primary data collection over the study period while South Africa (University of Witwatersrand Medical School) will provide secondary data consisting of a minimal dataset and relevant collected samples for analysis. All these centers have existing diabetes care clinics with experienced staff who are used to collecting and providing data for research purposes.

Eligibility: All patients with a clinical diagnosis of type 1 diabetes or young-onset insulin treated diabetes, who were diagnosed before the age of 30 years will be eligible to be enrolled into the study. We estimated a minimum total sample size of 500 participants will have a high precision with 95% confidence intervals of 17-25% around a prevalence of 20% for a clinical or biological characteristics (e.g. retained C-peptide or presence of islet auto-antibodies) and 46-54% around a prevalence of 50%.

Sampling method: We will follow a systematic sampling method, enrolling consecutive eligible participants from the different primary collection clinical sites.

Enrollment: All consented patients will be interviewed using a structured pre-tested questionnaire (Data Collection Form) by a trained study staff to collect relevant information; demographic, socioeconomic, lifestyle, family history, history of diabetes and diabetes complications. The questionnaire used in this study is available in English and has been translated into the major local language(s); the appropriate questionnaire is used according to the participant's preference. After the interview, a short clinical examination will be performed to record anthropometric characteristics (weight, height, waist and hip circumferences) and blood pressure.

Using standardized operating procedures (SOPs), saliva, blood and urine samples will be collected from all study participants for biochemical analysis, and biobanking for future studies. Saliva will be used for DNA extraction and for the determination of type 1 genetic risk score (T1D GRS) using a 67 single nucleotide polymorphism score as described by Sharp et al. 2019. Venous whole blood will be used for full blood count and A1c determination. Plasma will be used for random C-peptide determination on the 801 module of the Cobas 8000 analyser and the measuring range will be truncated to <3pmol/L. Serum creatinine will be measured to assist in the interpretation of the C-peptide result. Islet autoantibodies, GAD, IA2 and ZnT8 will be measured in serum on the RSR Limited ELISA (RSR Limited, Cardiff, U.K.). Dipstick urinalysis will be done, with urinary C-peptide and creatinine measurement for the determination of the urinary C-peptide to creatinine ration (UCPCR). .

Data collected from the different clinical sites using the data collection form will be entered into a centralized data management tool (REDCap). All data will be anonymised before being stored in the data management system.

Ethical consideration: All participants will be required to provide a written informed consent before participating in the study. Refusal to participate will not affect the quality of care of the participants at the clinical sites. The study has received ethical clearance from the National Ethics Committee of Cameroon ( No 2018/12/1252/L/CNERSH/SP), and the Uganda Virus Research Institute (GC/127/19/12/736), Muhimbili National Hospital (MNH/IRB/I/2020/019) and Human Research Ethics Committe, South Africa (M200174).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes at age less than 30 years
* Currently use insulin as a permanent treatment
* Able to consent to study

Exclusion Criteria:

* Refusal to provide written informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population is patients with clinically diagnosed type 1 diabetes or diagnosed with young-onset diabetes who are on permanent insulin therapy and being followed-up at the selected different clinical sites across the three countries. The diagnosis of diabetes must have been made before the age of 30 years.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of retained endogenous insulin secretion | Baseline
  Random non-fasting C-peptide level
Islet auto-antibody titre and positivity proportions | Baseline
  GADA, IA-2A, ZnT8A

SECONDARY OUTCOMES:
Type 1 diabetes genetic risk score | Baseline
  Proportion with T1D GRS > 50th centile

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sobgnwi, MD, PhD, Principal Investigator — University of Yaounde 1/ Yaounde Central Hospital
Locations (4):
- National Obesity Centre, Yaounde Central Hospital, Yaoundé, Centre Region, Cameroon
- School of Pathology, University of Witwatersrand, Johannesburg, Gauteng, South Africa
- Muhimbili National Hospital, Dar es Salaam, Tanzania
- Uganda Virus Research Institute, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Yes
A data sharing plan has been developed and validated by all the institutions. All data produced will be anonymized at the clinical site based on pre-existing data codes that have been generated. The data will be kept at a central data hub with all individual principal researchers having access to the data. The data produced during the course of study can be shared upon reasonable request to the Global Health Research Group study committee.
Supporting Information: Study Protocol, SAP
Time Frame: All data produced during the course of the study are entered and held at the central data management hub with access to all principal study investigators in real time as they are uploaded into the system. The data will be held on the server up to 5 years after the closure of recruitment in 2022.
Access Criteria: Access to the main data hub which is being controlled by the Global Health Research Group at the University of Exeter will be granted to country principal investigators who can remotely access the database from their different locations with their personal secured credentials.
URL: https://universityofexeteruk.sharepoint.com/sites/GlobalHealthDiabetesResearch/

REFERENCES:
- [Background] Sharp SA, Rich SS, Wood AR, Jones SE, Beaumont RN, Harrison JW, Schneider DA, Locke JM, Tyrrell J, Weedon MN, Hagopian WA, Oram RA. Development and Standardization of an Improved Type 1 Diabetes Genetic Risk Score for Use in Newborn Screening and Incident Diagnosis. Diabetes Care. 2019 Feb;42(2):200-207. doi: 10.2337/dc18-1785. PMID 30655379